CLINICAL TRIAL: NCT01780662
Title: A Phase 1/2 Study of Brentuximab Vedotin (SGN35) in Combination With Gemcitabine for Pediatric and Young Adult Patients With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin and Gemcitabine Hydrochloride in Treating Younger Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00107; NCI-2013-00107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AHOD1221; COG-AHOD1221; AHOD1221 (Other: Children's Oncology Group); AHOD1221 (Other: CTEP); U10CA180886 (NIH); UM1CA097452 (NIH)
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Recurrent Adult Hodgkin Lymphoma; Recurrent Childhood Hodgkin Lymphoma; Refractory Childhood Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (brentuximab vedotin, gemcitabine hydrochloride) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on day 1 and gemcitabine hydrochloride IV over 100 minutes on days 1 and 8. Treatment repeats every 21 days for up to 15 more courses in the absence of disease progression or unacceptable toxicity. Patients with CR after any course may go off protocol therapy for stem cell transplant.
  Interventions: Drug: Brentuximab Vedotin; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011

SUMMARY:
This phase I/II trial studies the side effects and the best dose of brentuximab vedotin when given together with gemcitabine hydrochloride and to see how well they work in treating younger patients with Hodgkin lymphoma that has returned or does not respond to treatment. Monoclonal antibodies, such as brentuximab vedotin, may find cancer cells and help kill them. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving brentuximab vedotin together with gemcitabine hydrochloride may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended Phase 2 dose of brentuximab vedotin in combination with gemcitabine administered every three weeks to children with relapsed or primary refractory Hodgkin lymphoma (HL).

II. To define and describe the toxicities of brentuximab vedotin in combination with gemcitabine administered on this schedule.

III. To determine the complete response (CR) rate after treatment with four cycles of gemcitabine with brentuximab vedotin among patients with relapsed or refractory HL.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of brentuximab vedotin in combination with gemcitabine within the confines of a Phase 1 study.

II. To describe the overall response rate (ORR) after 4 cycles of therapy among patients with relapsed or refractory HL.

III. To describe the proportion of patients with HL able to mobilize an adequate yield of cluster of differentiation (CD) 34+ stem cells after gemcitabine with brentuximab vedotin.

IV. To describe the relationship between disease response among patients with HL and changes in thymus and activation-regulated chemokine (TARC) during treatment, and to determine if specific micro ribonucleic acid (miRNA) profiles correlate with response to treatment.

V. To describe the frequency of the Fc gamma receptor IIIa (FcγRIIIa)-158 valine (V)/phenylalanine (F) polymorphism among patients who experience pulmonary toxicity on this protocol.

OUTLINE: This is a phase I, dose-escalation study of brentuximab vedotin followed by a phase II study. (Phase I completed as of amendment 4)

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1 and gemcitabine hydrochloride IV over 100 minutes on days 1 and 8. Treatment repeats every 21 days for up to 15 more courses in the absence of disease progression or unacceptable toxicity. Patients with CR after any course may go off protocol therapy for stem cell transplant.

After completion of study treatment, patients are followed up at 3, 6, 9, 12, 18, 24, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of the malignancy at original diagnosis; patients must have histologic verification of recurrent Hodgkin disease at the time of relapse; no additional biopsy is required for patients with primary refractory disease (i.e. no prior CR)
* PARTS A AND B: Patients with Hodgkin lymphoma (HL) are eligible for both the phase 1 and 2 portions, if they are in one of the following categories:

  * Primary refractory disease (i.e. no prior CR)
  * Very early relapse (< 6 months from the end of initial therapy, including chemotherapy ± radiation)
  * Advanced stage (III or IV) at diagnosis who relapse less than one year from the end of initial therapy
  * Note that patients with low-stage disease (IA or IIA) at initial diagnosis, who were treated with radiation alone or fewer than four cycles of chemotherapy will NOT be eligible
* Patients must have measurable disease, documented by clinical and radiographic criteria
* Patients must have a life expectancy of >= 8 weeks (>= 56 days)
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy

  * At least 14 days after the last dose of myelosuppressive chemotherapy (28 days if prior nitrosourea); Note: cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of therapy
  * At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * At least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
  * At least 3 half-lives of the antibody after the last dose of a monoclonal antibody
  * At least 14 days after local palliative radiation therapy (XRT) (small port); at least 150 days must have elapsed if prior total body irradiation (TBI), craniospinal XRT or if >= 50% radiation of pelvis; at least 42 days must have elapsed if other substantial bone marrow (BM) radiation
  * Patients with prior autologous or allogeneic stem cell transplant (SCT) are excluded from this study
  * At least 28 days must have elapsed since the most recent dose of bleomycin, to allow adequate time to detect evidence of bleomycin-related pulmonary toxicity
* PART A: FOR PATIENTS WITH KNOWN BONE MARROW INVOLVEMENT (Completed as of Amendment 4)
* Peripheral absolute neutrophil count (ANC) >= 1000/uL
* Platelet count >= 100,000/uL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* PART B: FOR PATIENTS WITHOUT KNOWN BONE MARROW INVOLVEMENT
* Peripheral absolute neutrophil count (ANC) >= 750/uL
* Platelet count >= 75,000/uL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with lymphoma metastatic to bone marrow who have granulocytopenia, anemia, and/or thrombocytopenia will be eligible for study but not evaluable for hematologic toxicity (in Part A, there will be a maximum of one per cohort); such patients must meet the blood counts as in Part A (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled in Part A must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 OR
* A serum creatinine based on age/gender as follows:

  * =< 0.6 mg/dL (for 1 to < 2 years of age)
  * =< 0.8 mg/dL (for 2 to < 6 years of age)
  * =< 1.0 mg/dL (for 6 to < 10 years of age)
  * =< 1.2 mg/dL (for 10 to < 13 years of age)
  * =< 1.4 mg/dL (for females >= 13 years of age)
  * =< 1.5 mg/dL (for males 13 to < 16 years of age)
  * =< 1.7 mg/dL (for males >= 16 years of age)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x upper limit of normal (ULN) for age; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* No evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and a pulse oximetry > 92% while breathing room air
* Forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) > 60% by pulmonary function test (PFT), unless due to large mediastinal mass from HL; carbon monoxide diffusion capacity (DLCO), FEV1, and forced vital capacity all > 50% predicted value; Note: pulmonary function testing is not required for children < 8 years old, or for any child who is developmentally unable to comply with pulmonary function testing
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4) resulting from prior therapy must be < grade 2

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during protocol therapy and for at least 30 days after the last dose of brentuximab vedotin; abstinence is an acceptable method of birth control
* Concomitant medications

  * Patients receiving stable or decreasing corticosteroids are not eligible for other concurrent conditions (e.g. asthma, autoimmune diseases, rash, documented adrenal insufficiency) are eligible for this study
  * Patients who are currently receiving another investigational drug are not eligible
  * Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients with an immunodeficiency that existed prior to diagnosis, such as primary immunodeficiency syndromes, organ transplant recipients and children on current systemic immunosuppressive agents are not eligible
* Patients known to be positive for human immunodeficiency virus (HIV) are not eligible
* Prior therapy

  * Patients with prior exposure to brentuximab vedotin are not eligible; NOTE: prior exposure to gemcitabine is NOT an exclusion criterion
  * Patients who have undergone prior autologous or allogeneic SCT are not eligible
  * Patients with HL who were stage IA or IIA at initial diagnosis and treated with either radiation alone or < 4 cycles of chemotherapy are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients with known hypersensitivity to Escherichia coli (E.coli)-derived proteins, filgrastim, or any component of filgrastim are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 13 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2013-01-31 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Cole, Principal Investigator — Children's Oncology Group
Locations (116):
- United States (109):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec

REFERENCES:
- [Derived] Cole PD, McCarten KM, Pei Q, Spira M, Metzger ML, Drachtman RA, Horton TM, Bush R, Blaney SM, Weigel BJ, Kelly KM. Brentuximab vedotin with gemcitabine for paediatric and young adult patients with relapsed or refractory Hodgkin's lymphoma (AHOD1221): a Children's Oncology Group, multicentre single-arm, phase 1-2 trial. Lancet Oncol. 2018 Sep;19(9):1229-1238. doi: 10.1016/S1470-2045(18)30426-1. Epub 2018 Aug 16. PMID 30122620

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a Phase I /II study. Phase I determined the Maximum Tolerated Dose (MTD) between the first 2 treatment arms; 16 patients enrolled and 9 patients completed therapy. The study was closed and reopened to accrual for Phase II which enrolled an additional 30 patients. Overall, 46 patients were enrolled but only 29 patients completed therapy.
Groups:
- Phase I, 1.4mg/kg: Patients who were enrolled in Phase I and took dose 1.4mg/kg
- Phase I, 1.8mg/kg: Patients who were enrolled in Phase I and took dose 1.8mg/kg
- Phase II, 1.8mg/kg: Patients who were enrolled in Phase lI and took dose 1.8mg/kg
Period: Overall Study
Arm/Group | Phase I, 1.4mg/kg | Phase I, 1.8mg/kg | Phase II, 1.8mg/kg
Started | 3 | 13 | 30
Completed | 2 | 7 | 20
Not Completed | 1 | 6 | 10
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Physician Decision | 0 | 5 | 7
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Ineligible | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I Dose 1.4 mg/kg: Patients who were enrolled in Phase I and took dose 1.4mg/kg
- Phase I Dose 1.8 mg/kg: Patients who were enrolled in Phase I and took dose 1.8mg/kg
- Phase 2 Dose 1.8 mg/kg: Patients who were enrolled in Phase lI and took dose 1.8mg/kg
- Total: Total of all reporting groups
Arm/Group | Phase I Dose 1.4 mg/kg | Phase I Dose 1.8 mg/kg | Phase 2 Dose 1.8 mg/kg | Total
Number analyzed (Participants) | 3 | 13 | 30 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 10 | 24 | 37
  Between 18 and 65 years | 0 | 3 | 6 | 9
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 16 | 25
  Male | 2 | 5 | 14 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 9 | 11
  Not Hispanic or Latino | 3 | 11 | 20 | 34
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 6 | 8
  White | 3 | 10 | 19 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 13 | 28 | 44
  Canada | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) for Brentuximab Vedotin
Description: MTD was determined as the maximum dose at which fewer than one-third of patients experience Dose Limiting Toxicities (DLT) as assessed by National Cancer Institute (NCI) CTCAE v 4.0 during Cycle 1 of therapy. Gemcitabine was administered on days 1 and 8 of a 21 day cycle at a fixed dose. Brentuximab vedotin was investigated at a starting dose of 1.4 mg/kg administered on day 1 and escalated if tolerated.
Time Frame: During cycle 1 of protocol therapy (21 days)
Population: The first 9 out of 16 patients enrolled with relapsed/refractory HL in a phase 1 dose finding study of brentuximab vedotin in combination with gemcitabine, were used in determining MTD
Measure: Number; unit: mg/kg
Arm/Group | Treatment (Brentuximab Vedotin, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 9
mg/kg | 1.8

2. Primary Outcome: Adverse Events Graded According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: The number of eligible patients assigned to receive brentuximab vedotin in combination with gemcitabine that experienced CTC Version 4, grade 3 or higher adverse events during Phase 1 and Phase 2.
Time Frame: 13 months from first dose
Population: All eligible patients (N=45). One patient was ineligible due to exceeding the prescribed interval between disease evaluation and study entry.
Measure: Count of Participants; unit: Participants
Groups:
- Dose 1.4mg/kg (Phase I): Patients who were enrolled in Phase I and took dose 1.4mg/kg
- Dose 1.8mg/kg (Phase I + Phase II): Patients who were enrolled in Phase I and Phase II and took dose 1.8mg/kg
Arm/Group | Dose 1.4mg/kg (Phase I) | Dose 1.8mg/kg (Phase I + Phase II)
Number analyzed (Participants) | 3 | 42
Participants
  Abdominal pain | 0 | 1
  Adrenal insufficiency | 0 | 1
  Alanine aminotransferase increased | 1 | 13
  Anemia | 1 | 4
  Anorexia | 0 | 1
  Aspartate aminotransferase increased | 1 | 10
  Dehydration | 0 | 1
  Dental caries | 0 | 1
  Diarrhea | 0 | 3
  Febrile neutropenia | 0 | 2
  GGT increased | 0 | 1
  Hemolytic uremic syndrome | 0 | 1
  Hypophosphatemia | 0 | 2
  Hypotension | 0 | 4
  Infections and infestations - Other- Specify | 0 | 1
  Investigations - Other- Specify | 0 | 1
  Lung infection | 0 | 2
  Lymphocyte count decreased | 3 | 8
  Myositis | 0 | 1
  Nausea | 0 | 2
  Neutrophil count decreased | 3 | 28
  Non-cardiac chest pain | 0 | 1
  Pain in extremity | 0 | 1
  Pericardial effusion | 0 | 1
  Platelet count decreased | 0 | 13
  Pneumonitis | 1 | 0
  Pruritus | 1 | 0
  Rash maculo-papular | 0 | 3
  Skin infection | 0 | 1
  Urinary tract infection | 0 | 1
  White blood cell decreased | 3 | 15

3. Primary Outcome: The Number of Patients With Relapsed or Refractory HL Who Achieved Complete Response (CR)
Description: The number of patients who experienced complete Response (CR) within the first four cycles. By modern response criteria, those with partial response (PR) or stable disease with all target lesions with Deauville scores <=3 after cycle 4 are also considered as CR. Patients were assessed after treatment with four cycles of gemcitabine with brentuximab vedotin. CR was only reported for Dose level 2 across both phases of study.
Time Frame: After 4 cycles (21 days per cycle) of protocol therapy
Population: All eligible patients (N=42) at Dose Level 2 (brentuximab vedotin 1.8 mg/kg with gemcitabine). 4 patients were excluded. 3 patients did not receive dose level 2 and 1 patient was ineligible due to exceeding the prescribed interval between disease evaluation and study entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Brentuximab Vedotin, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 42
Participants | 28

4. Secondary Outcome: The Number of Patients Who Had Disease Response Assessed by Deauville Scales Among Those in Phase I With Dose Level 2.
Description: The Deauville five-point scale was used to assess the number of participants with complete response (CR) and partial response (PR). A lower score indicates a better outcome. Scores of 1-3 represent CR and 4-5 represent PR.
Time Frame: Up to 13 months from first dose
Population: All eligible patients in phase 1, dose level 2 (N=13). 3 patients in phase 1 were not given dose level 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Brentuximab Vedotin, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 13
Participants | 8

5. Secondary Outcome: Percentage of Patients Who Achieved Overall Response (OR) as Measured by Complete Response (CR) and Partial Response (PR)
Description: The percentage of patients who experienced complete Response (CR) within the first four cycles.By modern response criteria, those with partial response (PR) or stable disease with all target lesions with Deauville scores <=3 after cycle 4 are also considered as CR. Patients were assessed after treatment with four cycles of gemcitabine with brentuximab vedotin. CR was only reported for Dose level 2 across both phases of study.
Time Frame: After 4 cycles (21 days per cycle) of protocol therapy
Population: All eligible patients (N=42) at Dose Level 2 (brentuximab vedotin 1.8 mg/kg with gemcitabine).4 patients were excluded. 3 patients did not receive dose level 2 and 1 patient was ineligible due to exceeding the prescribed interval between disease evaluation and study entry.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Brentuximab Vedotin, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 42
percentage of participants | 74 [58 to 86]

6. Secondary Outcome: The Number of Patients Who Had Successful Peripheral Blood Stem Cell (PBSC) Collection
Description: Successful PBSC collection was defined as a collection of more than 2x10^6 CD34 positive cells.
Time Frame: From 1 to 5 cycles
Population: For 21 of the eligible 45 subjects, PBSC collection was not attempted during protocol therapy, either because stem cells had been collected prior to study enrollment, or no autologous stem cell transplant was planned. 1 patient was ineligible due to exceeding the prescribed interval between disease evaluation and study entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Brentuximab Vedotin, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 24
Participants | 24

7. Secondary Outcome: Plasma Level of Thymus and Activation-Regulated Chemokine (TARC)
Description: Limit to 41 evaluable patients who received dose 1.8 mg/kg
Time Frame: From baseline to time prior to cycle 2
Population: 4 eligible patients did not consent for genetic studies. 3 of the 41 did not have baseline TARC and 6 did not have TARC prior to cycle 2.
Measure: Median (Full Range); unit: pg/ml
Groups:
- Dose 1.8mg/kg: Evaluable patients who received dose 1.8mg/kg.
Arm/Group | Dose 1.8mg/kg
Number analyzed (Participants) | 41
pg/ml
  Baseline: number analyzed (Participants) | 38
  Baseline | 5700 [389 to 18,667]
  Prior to Cycle 2: number analyzed (Participants) | 35
  Prior to Cycle 2 | 668 [6 to 9,718]

8. Secondary Outcome: Correlation Between Micro Ribonucleic Acid (miRNA) and Disease Response to Protocol Treatment
Description: Limit to 41 evaluable patients who received dose 1.8 mg/kg
Time Frame: From the end of first dose to the end of last dose (Up to 13 Months)
Population: These samples were banked but not analyzed, due to a change in research priorities.
Arm/Group | Treatment (Brentuximab Vedotin, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Patients With FcyRIIIa-158 V/F (Valine/Phenylalanine) Polymorphism
Description: Among patients who received 1.8mg/kg dose, the frequency of the FcγRIIIa-158 V/F polymorphism are described.
Time Frame: From the end of first dose to the end of last dose (Up to 13 Months)
Population: 4 eligible patients did not consent for genetic studies.
Measure: Count of Participants; unit: Participants
Groups:
- Dose 1.8mg/kg: Evaluable patients with received dose of 1.8mg/kg
Arm/Group | Dose 1.8mg/kg
Number analyzed (Participants) | 41
Participants
  Homozygous FF- Phenylalanine | 22
  Heterozygous FV- Valine/Phenylalanine | 14
  Homozygous VV- Valine | 5

ADVERSE EVENTS:
Time Frame: From first dose up to 13 months.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Groups:
- Dose1.4mg/kg; Dose 1.8mg/kg: Patients receive brentuximab vedotin IV over 30 minutes on day 1 and gemcitabine hydrochloride IV over 100 minutes on days 1 and 8. Treatment repeats every 21 days for up to 15 more courses in the absence of disease progression or unacceptable toxicity. Patients with CR after any course may go off protocol therapy for stem cell transplant.
  Brentuximab Vedotin: Given IV
  Gemcitabine Hydrochloride: Given IV
Arm/Group | Dose1.4mg/kg | Dose 1.8mg/kg
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/42
Serious Adverse Events (participants affected / at risk) | 3/3 | 37/42
Other Adverse Events (participants affected / at risk) | 3/3 | 28/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose1.4mg/kg (N=3) | Dose 1.8mg/kg (N=42)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Infections and infestations - Other- Specify (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 13 (13)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 10 (10)
GGT increased (Investigations) | 0 (0) | 1 (1)
Investigations - Other- Specify (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (3) | 8 (8)
Neutrophil count decreased (Investigations) | 3 (3) | 28 (28)
Platelet count decreased (Investigations) | 0 (0) | 13 (13)
White blood cell decreased (Investigations) | 3 (3) | 15 (15)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose1.4mg/kg (N=3) | Dose 1.8mg/kg (N=42)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 6 (6)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ear and labyrinth disorders - Other- Specify (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 9 (9)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 8 (8)
Chills (General disorders) | 0 (0) | 2 (2)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 8 (8)
Fever (General disorders) | 1 (1) | 8 (8)
General disorders and administration site conditions - Other- Specify (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Phlebitis infective (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 9 (9)
Alkaline phosphatase increased (Investigations) | 0 (0) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 10 (10)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Carbon monoxide diffusing capacity decreased (Investigations) | 0 (0) | 2 (2)
CPK increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Investigations - Other- Specify (Investigations) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (4)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 5 (5)
Weight gain (Investigations) | 2 (2) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 7 (7)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other- Specify (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory- thoracic and mediastinal disorders - Other- Specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 12 (12)
Skin and subcutaneous tissue disorders - Other- Specify (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Surgical and medical procedures - Other- Specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Samples have been banked, but data will never be analyzed for Outcome measure #8, Correlation between micro ribonucleic acid (miRNA) and disease response to protocol treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT01780662/Prot_SAP_000.pdf